CLINICAL TRIAL: NCT00000996
Title: Phase II Study of Weekly Doxorubicin Treatment of AIDS Associated Kaposi's Sarcoma
Brief Title: A Study of Doxorubicin in the Treatment of AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 006; 10982 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Doxorubicin; Drug Evaluation; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin hydrochloride

SUMMARY:
To study the natural course of AIDS related Kaposi's sarcoma and to determine the usefulness and safety of weekly administration of small doses of doxorubicin.

Doxorubicin is one of the most active of all antitumor agents but at currently used doses toxicity is common. When small doses are administered on a weekly schedule, the toxicity of the drug appears to be reduced.

DETAILED DESCRIPTION:
Doxorubicin is one of the most active of all antitumor agents but at currently used doses toxicity is common. When small doses are administered on a weekly schedule, the toxicity of the drug appears to be reduced.

Patients are stratified for non-therapy purposes into 2 groups; doxorubicin is given intravenously (IV) every week on an outpatient basis. Patients are monitored carefully, and weekly blood samples are taken to determine the effectiveness and safety of treatment. Patients are evaluated for toxicity after one dose of the drug and weekly thereafter. Patients are evaluated for response to the drug after 4 weeks and monthly thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Ongoing and/or maintenance therapy for opportunistic infection.
* Medications for nausea, vomiting, and diarrhea resulting from drug.

Patients must have AIDS related Kaposi's sarcoma.

* Patients may demonstrate positive blood cultures for Mycobacterium avium-complex or cytomegalovirus.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions will be excluded:

* Patients with active opportunistic infection.
* Patients with concurrent neoplasm other than squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
* Patients with significant neurologic, cardiac, or liver disease.

Concurrent Medication:

Excluded:

* Antiretroviral agents.
* Immunomodulators.
* Corticosteroids.
* Experimental drugs.

The following patients will be excluded from the study:

* Patients with lymphadenopathy alone and/or visceral disease alone secondary to Kaposi's sarcoma.

Prior Medication:

Excluded:

* Cytotoxic chemotherapy.
* Excluded within 30 days of study entry:
* Antiretroviral agents.
* Biologic modifiers.
* Corticosteroids.

Prior Treatment:

Excluded:

* Total body electron beam therapy.
* Excluded within 30 days of study entry:
* Radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Study Completion 1990-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MA Fischl, Study Chair
Locations (12):
- United States (12):
  - UCLA CARE Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio

REFERENCES:
- [Background] Walker RE, et al. The safety, pharmacokinetics, and antiviral activity of N-acetylcysteine in HIV-infected individuals. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo8 (abstract no MoB 0022)
- [Background] Fischl MA, Krown SE, O'Boyle KP, Mitsuyasu R, Miles S, Wernz JC, Volberding PA, Kahn J, Groopman JE, Feinberg J, et al. Weekly doxorubicin in the treatment of patients with AIDS-related Kaposi's sarcoma. AIDS Clinical Trials Group. J Acquir Immune Defic Syndr (1988). 1993 Mar;6(3):259-64. PMID 8450401